CLINICAL TRIAL: NCT06650943
Title: Efficacy Study on Nursing Consultation in Weight and Metabolic Syndrome Management Based on the Carbohydrate-insulin Theory in Individuals with First-episode Psychosis (MetaKOP)
Brief Title: Nursing Intervention in Weight and Metabolic Syndrome Management in First-episode Psychosis (MetaKOP)
Acronym: MetaKOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Basurto (Other)
Collaborators: Euskal Herriko Unibertsitatea. Universidad del Pais Vasco. (Unknown); Instituto Vasco de InvestigaciÃ³n Sanitaria (BIOEF) (Unknown)
Responsible Party: Principal Investigator, Lander Madaria Marijuan, Mental Health Nurse Specialist, Hospital de Basurto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 48.23 CEIHU
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: First Episode Psychosis (FEP); Metabolic Syndrome X
Keywords: FEP; psychosis; metabolic syndrome; nursing; mental health nurse
MeSH Terms: conditions — Metabolic Syndrome; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The psychometric scale evaluators will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention consists of 8 nursing consultations with a mental health nurse trained in healthy habits for individuals with psychosis. During the first 2 months, 4 consultations will focus on dietary habits based on the carbohydrate-insulin theory and physical activity, following a guide developed by experts, incorporating recommendations from the American Diabetes Association. Visits 5 and 6 occur at 3 and 4 months; visit 7 at 6 months to evaluate effectiveness, and visit 8 at 12 months. Weight will be monitored throughout. Assessments at baseline, 6, and 12 months will include labs, vital signs, and scales for psychopathology, quality of life, and activity level. Each session covers key topics, from intervention goals to diet tips and physical activity. The approach is flexible, aiming for gradual habit integration, supported by a therapeutic relationship. Phone reminders will enhance adherence.
  Interventions: Behavioral: Nursing Consultation in Weight Management and Metabolic syndrome
- Control (No Intervention): Ccontrol group will continue their usual follow-up within the EIP, attending consultations with their reference psychiatrist and receiving pharmacological or psychotherapeutic treatment as they did before the intervention. The control group will not receive any specific nursing consultations (beyond the administration of long-acting injectable antipsychotics where appropriate) or dietary or lifestyle advice during the follow-up. If patients in the control group require treatment or assistance for metabolic problems, they will be referred to primary care or endocrinology professionals, as was done previous to the intervention implementation.

INTERVENTIONS:
Behavioral: Nursing Consultation in Weight Management and Metabolic syndrome — Based on the Carbohydrate-insulin Theory
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to evaluate if a nursing intervention based on the carbohydrate-insulin model can effectively reduce weight and manage the risk of metabolic syndrome (MetS) in individuals with first-episode psychosis. The main questions it aims to answer are:

Will the intervention lead to a clinically significant weight loss (≥5%)? Can the intervention improve metabolic parameters, psychopathological state, physical activity level, and quality of life? Researchers will compare participants receiving the specialized nursing consultations to those receiving routine care to see if the former group experiences greater improvements in weight loss and metabolic risk reduction.

Participants will:

Attend a series of 8 nursing consultations focused on dietary habits based on the carbohydrate-insulin model and physical activity.

Complete assessments at the start, 6 months, and 12 months, including weight, metabolic parameters, and psychological evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to the Early Intervention Program (EIP).
2. First-episode psychosis (FEP) within the last 5 years.
3. Diagnosis of psychosis from the F2 spectrum or an affective disorder with psychotic symptoms according to ICD-10.

Exclusion Criteria:

1. Cognitive inability to learn or comorbid intellectual disability that interferes with study procedures.
2. Comorbid diagnosis of neurological pathology.
3. Language or comprehension impairments preventing accurate data collection.
4. Use of hypoglycemic medication before or during the study.
5. Refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Weight | From enrollment to the end of treatment at 48 weeks
  Weight in kilograms

SECONDARY OUTCOMES:
Metabolic Syndrome | From enrollment to the end of treatment at 48 weeks
  According to the International Diabetes Federation (IDF)
Psychopathology | From enrollment to the end of treatment at 48 weeks
  measured using PANSS scale
Depressive symptoms | From enrollment to the end of treatment at 48 weeks
  measured by Hamilton Depression Rating Scale
Qualit of Life | From enrollment to the end of treatment at 48 weeks
  EuroQoL 5D scale will be used
Reported phisical activity | From enrollment to the end of treatment at 48 weeks
  International Physical Activity Questionnaire (IPAQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Basurto, Bilbao, Vizcaya, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madaria L, Aymerich C, Catalan A, Gonzalez-Torres MA. Protocol of an Efficacy Study on Nursing Consultation in Weight Management and Metabolic Syndrome Based on the Carbohydrate-Insulin Theory in Individuals with First-Episode Psychosis. Nurs Rep. 2024 Dec 27;15(1):3. doi: 10.3390/nursrep15010003. PMID 39852625